CLINICAL TRIAL: NCT04124549
Title: Construction and Empirical Study of Exercise Program in Maintenance Hemodialysis Patients
Brief Title: The Effect of Intradialytic Combined Exercise on Physical Outcomes in End-Stage Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Mei Huang, student, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018538
Record Dates: First submitted 2019-09-25; First posted 2019-10-11 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Kidney Failure, Chronic; Exercise; Physical Fitness
Keywords: End-Stage Renal Disease; Exercise; Dialysis Efficacy; Physical Fitness
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients in the HD centers were randomly assigned to one of two wards at the time that they began to HD in this center. And in order to avoid contamination, randomization in this study was in accordance with the centers to which patients were assigned. Every HD center was randomized to either continue on usual HD care (control group) or intervention of intradialytic combined exercise based on usual HD care (intervention group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stand of Care (Sham Comparator): Patients in the control group received usual care with sham exercise.
  Interventions: Other: Usual care with sham intervention
- Combined Exercise (Experimental): The intervention was a 24-week progressive intradialytic combined cycling exercise which proceed in the first HD 2 hours. Each exercise lasted about 40 minutes.
  Interventions: Other: Intradialytic Combined Exercise

INTERVENTIONS:
Other: Usual care with sham intervention — Patients in the control group received usual care and were advised to do sham exercise such as stretch legs and arms about 15 minutes during the first 2 HD hours.
  Arms: Stand of Care
Other: Intradialytic Combined Exercise — Each session consisted of a 5-minute warm-up, cool-down and 30-minute cycling at a Rating of Perceived Exertion (RPE) of 12-14. The machine has two exercise types including aerobic exercise and resistance exercise. Patients were asked to perform aerobic exercise 20-min and resistance exercise 10-min in the first stage. Every four weeks is divided into a stage. And the time of aerobic exercise and resistance exercise were personally adjusted per stage to maintain the personalized target RPE. In the following stages, aerobic exercise was continued 15-min for the second stage, 10-min for the third and the forth stage, 15-min for the fifth stage and 20-min for the last stage. And the time for resistance exercise was adjusted for the total exercise time. The resistance of exercise also progressive increased in order to adapt the target RPE. It was accessible to patients of different ages, gender, cultures and ethnicities.
  Arms: Combined Exercise

SUMMARY:
Hemodialysis (HD) is an important and commonly used renal replacement therapy (RRT) for End-Stage Renal Disease (ESRD) patients worldwide. Inadequate HD, impaired exercise capacity and declined peripheral muscular strength resulted by HD and ESRD are still disturbing problems, which also predicts poor renal prognosis and poor quality of life. The results of systematic reviews by the investigators have shown that aerobic exercise and combined exercise can improve dialysis efficacy (alleviate uremia symptoms), improve aerobic exercise capacity and muscle strength, and improve patients' quality of life, which also supports the notion that the National Kidney Foundation Disease Outcomes Quality Initiative (K/DOQI) recommends exercise as cornerstone of ESRD rehabilitation. Therefore, this study used the effective exercise type of the systematic review results - combined exercise as an intervention method to observe its effects on dialysis efficacy, blood pressure, aerobic exercise capacity, muscle strength and quality of life.

The study hypothesized that combined exercise can not only improve dialysis efficacy, but also has an interaction effect with intervention duration, which deserves researches' attention. Combined exercise will also improve blood pressure (including systolic blood pressure and diastolic blood pressure) in patients with ESRD and reduce the symptoms of renal hypertension. It will also improve the exercise capacity and muscle strength of ESRD patients and improve their quality of life.

DETAILED DESCRIPTION:
Hemodialysis (HD) is an important and commonly used renal replacement therapy (RRT) for End-Stage Renal Disease (ESRD) patients worldwide. Single-pool Kt/V (sp Kt/V) is a quantified indicator of HD adequacy and has been recommended should be more than 1.2 by The National Kidney Foundation Disease Outcomes Quality Initiative (K/DOQI). Inadequate HD predicted increased hospitalization time and cost and reduced survival time. Increasing dose or frequency were common clinical therapies to improve HD adequacy but were limited by patients' poor compliance and greater finical burden. Economical and affordable methods to increase urea and other toxins are urgent clinically.

Physical fitness decline, often accompanied with sedentary lifestyle are also disturbing issues for ESRD. And physical fitness reduction would exacerbate with the extension of HD years. In addition, patients should sit or lie still for 4 hours during HD and post-dialysis fatigue worsened physical function. Exercise capacity and peripheral muscular strength had 40% to 50% reduction compared to same age and gender, which resulted from metabolic disorders and physiological deterioration of HD. Then muscle functionality and cardiorespiratory capacity declined and reflected in reduction of physical function which was a risk factor of poor renal prognosis and poor quality of life.

Exercise was an economical way and was recommended by K/DOQI as cornerstone of rehabilitation for HD patients. There are kinds of exercise intervention, including aerobic exercise, resistance exercise and aerobic and resistance exercise (combined exercise), which showed obvious beneficial effects on the recovery for HD patients, such as mitigating patients' uremic symptoms, elevating their physical fitness and improving quality of life (QoL) in recent 30 years' studies. Previous studies showed that sp Kt/V can be elevated not only by single exercise intervention, but also by long term intervention. But there are few studies observed the interaction between time and exercise in the long term exercise intervention. About physical fitness, exercise, especially aerobic exercise, can increase patients' aerobic capacity, such as maximal peak oxygen and walking ability. Exercise also has a marked effect on muscle strength, with resistance exercise reducing muscle wasting and enhancing muscle strength.

According to the investigators' previous meta-analysis, both aerobic exercise and combined exercise can increase patients' exercise capacity and QoL. Investigators prefer choosing combined exercise because few researches regard combined exercise as intervention exercise type which can provide more information to future systematic reviews. About the exercise time, investigators chose intradialytic exercise for good compliance, professional guidance and clinical professional guarantee. As for the duration, intensity and frequency, 6 months, moderate intensity and 3 times per week may good for restore blood vessel structure, physical function and quality of life from the investigator's previous result. Above all, this study aimed to invest the effect of intradialytic combined exercise on sp Kt/V, walking ability, muscle strength and QoL.

The randomized, parallel-controlled trial aimed to compare the effect of 24 weeks combined exercise and usual care on hemodialysis efficacy, functional capacity and quality of life in patients with ESRD on HD. The protocol of this study was conducted in accordance with the Declaration of Helsinki and was reviewed and approved by the Human Research Ethics Committee of the Xi'an Jiaotong University Health Science Center (No 2018538), China. Informed consent was obtained from participants in this study.

Data analysis Continuous data were expressed as mean and standard deviation (SD) or median and interquartile range according to the normality results. Proportion data were expressed as percentage frequency. The demographics of patient in two groups were compared. The Student T-test or Mann-Whitney U test where appropriate for the continuous data, and the Chi-square test was used for proportion data. The intragroup differences analysis was detected with the paired Student T-test or Wilcoxon rank test. Unpaired Student T-test or Mann-Whitney U test was evaluated the intergroup difference. In order to compare monthly data of sp Kt/V, two-way analysis of variance for repeated measures: group (presence or absence of intervention) and time (every 4 weeks) was performed. The differences were considered as statistical significant when P-values were ≤0.05. EpiData 3.1 (Odense, Denmark) was used for data entry, and the analyses were carried out using Statistical Product and Service Solutions (SPSS) 13.0 for Windows (Chicago, U.S.A).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age≥18) with stable ESRD.
* Receiving≥3 months HD.
* HD 3 times per week.
* Volunteer for participating this trial.

Exclusion Criteria:

* Unable to exercise (severe musculoskeletal pain at rest or with minimal activity precluding walking or stationary cycling; unable to sit, stand or walk unassisted) (walking device such as cane or walker allowed).
* Had shortness of breath at rest or with activities of daily living (NYHA Class IV).
* Had mental disease, disturbance of consciousness and couldn't cooperate with investigations and exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Dialysis Efficacy (sp Kt/V) | sp Kt/V was measured at baseline (before intervention) and after 24 weeks of intervention.
  Sp Kt/V is a dimensionless, mathematical representation of serum urea clearance, monitored by On-Line Clearance Monitor (OCM)-equipped Fresenius 4008-S machines (Fresenius, Bad Homburg, Germany).
Dialysis Efficacy (sp Kt/V) | sp Kt/V was measured after 4, 8, 12, 16 and 20 weeks of intervention for observing the effects of intervention and time on sp Kt/V more accurately.
  Sp Kt/V is a dimensionless, mathematical representation of serum urea clearance, monitored by On-Line Clearance Monitor (OCM)-equipped Fresenius 4008-S machines (Fresenius, Bad Homburg, Germany).

SECONDARY OUTCOMES:
Blood Pressure (including systolic blood pressure (SBP) and diastolic blood pressure (DBP)) | BP was measured at baseline (before intervention), 12 weeks after intervention and 24 weeks after intervention.
  were measured by the BP monitor of Fresenius 4008-S machines on the upper limb without arteriovenous fistula when the patients lay in the bed, ready to HD.
Six-minute walk test (6MWT) | 6MWT was measured at baseline (before intervention), 12 weeks after intervention and 24 weeks after intervention.
  6MWT is commonly used to assess walking capacity in patients with chronic diseases, including Chronic Kidney Disease (CKD) patients.
5-repetition sit-to-stand test (STS 5) | The STS-5 was measured at baseline (before intervention), 12 weeks after intervention and 24 weeks after intervention.
  The STS-5 were performed to measure lower extremity muscle capacity force.
30-second sit-to-stand test (STS 30) | The STS-30 was measured at baseline (before intervention), 12 weeks after intervention and 24 weeks after intervention.
  STS-30 were performed to measure lower extremity muscle capacity force
Kidney Disease Quality of Life (KDQOL-36) | The KDQOL-36TM was measured at baseline (before intervention), 12 weeks after intervention and 24 weeks after intervention.
  KDQOL-36, consisted of the 12-item Short Form Health Survey (SF-12) including the physical component summary (PCS) and the mental component summary (MCS) and 24 disease-specific items which entail 3 subscales: the symptom and problems list, the burden of kidney disease, and the effects of kidney disease, is to evaluate patients' QoL. Scores of each dimension range from 0 to 100 and higher scores represent better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Aili Lv, Doctor, Study Director — Xi'an Jiaotong University Health Science Center
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-11-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04124549/ICF_000.pdf